CLINICAL TRIAL: NCT03727412
Title: Post Implantation Syndrome and Administration on NSAIDs in Patients Undergoing Endovascular Repair of an Abdominal Aortic Aneurysm Under General Anesthesia
Brief Title: Post Implantation Syndrome and Administration on NSAIDs in Patients Undergoing EVAR for AAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Aneurysm Abdominal; Endovacular Repair
Keywords: post implantation syndrome; EVAR; cardiovascular outcome; NSAIDs
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Pharmaceutical Preparations; Drugs, Generic; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naproxen Group (Active Comparator): patients with an abdominal aortic aneurysm undergoing endovascular epair and taking preoperatively naproxen (Naprosyn, tab 500 mg twice/day for 4 days)
  Interventions: Drug: Drugs, Generic (Naprosyn)
- Control group (Placebo Comparator): patients with an abdominal aortic aneurysm undergoing endovascular epair and taking placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Drugs, Generic (Naprosyn) — naproxen administration perioperatively in patients with a abdominal aortic aneurysm undergoing endovascular repair
  Arms: Naproxen Group
Drug: Placebo Oral Tablet — placebo administration perioperatively in patients with a abdominal aortic aneurysm undergoing endovascular repair
  Arms: Control group

SUMMARY:
INTRODUCTION Post-implantation syndrome is the clinical and biochemical expression of an inflammatory response following endovascular repair of an aortic aneurysm. PIS is mainly a clinical condition associated with the implantation of an endograft and is diagnosed by the presence of fever accompanied by elevated WBC count above normal without any evidence of an infection.

The correlation between the type of the endograft placed and the development of PIS may indicate that the inflammatory reaction is due to the material of the endograft itself ( polyester or PTFE ). Based on the results of different studies the type of endograft's material seems to play an important role in PIS development and may have a predictive role for a significant number of patients undergoing endovascular repair of abdominal aortic aneurysm (EVAR).

In most studies PIS is considered a benign condition, although it may lead to a more demanding postoperative care characterized by prolonged hospitalization. In an other prospective study patients with PIS were more likely to suffer from an adverse event during the 30 days after the procedure. The occurrence of PIS was the only independent predictor of a MACE ( major cardiovascular events ) or an adverse event during the follow-up period.

Current available literature data certainly raise the question of altering current approach and treat patients with PIS by focusing on the reduction of the inflammatory response by administration of steroid or non-steroidal drugs.

The aim of the present randomized placebo-controlled study is to evaluate whether the perioperative administration of Naproxen (NPR) an anti-inflammatory drug with a beneficial cardiovascular safety profile in patients with an abdominal aortic aneurysm undergoing endovascular repair could have any effect on the inflammatory response and patients outcome during the first year of follow-up after the surgery.

METHOD PIS will be considered as the presence of fever (persisting body temperature > 38 ° C lasting more than 1 day during hospitalization) and leukocytosis ( white blood cell count > 12,000 / mL ) with negative blood and urine culture. All patients with AAA that will be subjected to EVAR in our department since February 2018 and who will receive an endograft made from polyester will be included in this study.

All patients after being informed pre-operatively about the way and the purpose of the clinical study, the patients will be randomly selected to receive either naproxen ( NPR ) 500 mg x 2 or placebo, starting the previous day before the procedure and for 3 days postoperatively. The NPR was selected due to the expected significant anti-inflammatory activity and favorable cardiovascular safety profile.

All patients presenting with fever during the post-operative period, whether or not fulfilling the PIS criteria, will undergo a thorough work up for possible infection. If any of these tests reveal evidence of an early pulmonary, urinary tract or any other kind of infection, the patient will not be considered to suffer from PIS. Patients will be discharged in the absence of any complications, with a body temperature < 38oC for at least 24 hours and a WBC < 12.000/mL.

Besides the traditional inflammatory markers (WBC, hs-CRP, and fibrinogen ) the investigators will also measure interleukin 6 (IL-6) because it was the only marker significantly altered in PIS patients in a previous study.

The follow-up will be performed at 1, and 12 months after surgery. Patient quality of life will also be studied by completing the SF36 questionnaire preoperatively and in the first year post-operative follow-up.

DETAILED DESCRIPTION:
INTRODUCTION Post-implantation syndrome is the clinical and biochemical expression of an inflammatory response following endovascular repair of an aortic aneurysm.1 PIS is mainly a clinical condition associated with the implantation of an endograft and is diagnosed by the presence of fever accompanied by elevated WBC count above normal without any evidence of an infection. The reported incidence of PIS in the literature has been varying widely from 14 to 60%.2-5 The correlation between the type of the endograft placed and the development of PIS may indicate that the inflammatory reaction is due to the material of the endograft itself (polyester or PTFE). Gerasimidis et al. in a relatively underpowered study concluded for the first time in 2005 that fever was more common in a group of patients receiving an endograft made from polyester in contrast to those receiving a PTFE graft. Interleukin 8 (IL-8) was higher in the first group, indicating a stronger host reaction in the specific material. Voute et al. in a later study showed that the implantation of stent grafts based on polyester was independently associated with a stronger inflammatory response. Moulakakis et al., observing a milder inflammatory activation in patients with a PTFE endograft, have confirmed this finding in a later report. Accordingly a previous study found that the use of polyester endograft independently predicted PIS and was correlated with an above 10 times higher risk for an inflammatory response. Based on the results of the above 3 mentioned studies the type of endograft's material seems to play an important role in PIS development and may have a predictive role for a significant number of patients undergoing endovascular repair of abdominal aortic aneurysm ( EVAR ).

The relation of PIS with patient's outcome has not been adequately established. In most studies PIS is considered a benign condition, although it may lead to a more demanding postoperative care characterized by prolonged hospitalization. In a prospective study of 214 patients after EVAR this group found that patients with PIS were more likely to suffer from an adverse event during the 30 days after the procedure. Adverse events occurred in 25.9% of the PIS group compared to 2.9% of the non- PIS group and included any major cardiovascular event, acute renal failure, readmission, and death by any cause. For the same cohort, at the 1-year follow-up, high-sensitivity C-reactive protein and interleukin 6 were attenuated toward the values of the non-PIS group. During the one-year follow-up period, MACE and adverse events occurred, respectively, in 17.2% and in 18.8% of patients in the PIS group and in 4.3% and 5.1% of the non-PIS group. The occurrence of PIS was the only independent predictor of a MACE or an adverse event during the follow-up period.

Current available literature data certainly raise the question of altering current therapeutic approach and treat patients with PIS by focusing on the reduction of the inflammatory response by administration of steroid or non-steroidal drugs. Motte et al published recently a prospective trial of 150 EVAR patients who were randomized to receive a single preoperative dose of methylprednisolone or placebo. The inflammatory response, as assessed by the inflammatory biomarkers levels, was reduced in the methylprednisolone group, although no differences were noted in patient outcomes between the two groups during a 3-month follow-up period. Data on postoperative use of anti-inflammatory drugs are absent.

Because PIS was the only independent predictor of an adverse event during the first year after EVAR, it seems that even a strong inflammatory stimulus at the immediate postoperative period could probably affect the cardiovascular health of these patients at the long term. Any therapeutic measurements that might thus focus on PIS acute treatment or even prevention seem reasonable.

The aim of the present randomized placebo-controlled study is to evaluate whether the perioperative administration of Naproxen (NPR) an anti-inflammatory drug with a beneficial cardiovascular safety profile17 in patients with an abdominal aortic aneurysm undergoing endovascular repair could have any effect on the inflammatory response and patients outcome during the first year of follow-up after surgery.

Patient quality of life will also be studied by completing the SF36 questionnaire preoperatively and in the first year post-operative follow-up.

METHOD According to the definition of PIS, it must fulfill at least two of the criteria of the Systemic Inflammatory Response Syndrome (SIRS), i.e. fever and leukocytosis. Therefore, PIS will be considered as the presence of fever (persisting body temperature > 38 ° C lasting more than 1 day during hospitalization) and leukocytosis ( white blood cell count > 12,000 / mL ) with negative blood and urine culture. All patients with AAA that will be subjected to EVAR from February 2018 and who will receive an endograft made from polyester will be included in this study.

Exclusion criteria will be clinical and / or laboratory indications of an infection preoperatively, including:

* Leukocytosis (white blood cell count [WBC]> 10,000 / mL) and elevated body temperature
* Signs of gangrene
* Previous trauma or surgery two months before enrolling in the study
* Previous implantation of endoprothesis
* Any autoimmune disease or systemic inflammatory condition
* Any malignancy
* Use of anti-inflammatory drugs, chemotherapeutic agents, immunosuppressants or anticoagulants
* Severe severe renal impairment (GFR < 30 ml / min) and
* Absolute contraindications of NSAIDs such as: NSAID-allergic patients, patients who have experienced asthma attacks following the use of acetylsalicylic acid or other anti-inflammatory nonsteroidal drugs, patients with nasal polyps, patients with anaphylactic or other severe NSAID allergies, severe hepatic insufficiency, heart failure patients (moderate to severe), patients with ischemic heart disease or other vascular diseases, presence of old or active gastric or ulcer of duodenum, history of gastrointestinal haemorrhage in the past, proctitis or recent rectal bleeding, a history of inflammatory bowel disease (ulcerative colitis, Crohn's disease).

After approval by the Scientific Council of the University Hospital of Larissa and written consent of all patients after being informed pre-operatively about the way and the purpose of the clinical study, the patients will be randomly selected to receive either Naproxen (NPR ) 500 mg x 2 or placebo, starting the previous day before the procedure and for 3 days postoperatively. The NPR has a half-life of 12-17 hours and reaches a maximum concentration at 1 to 4 hours after administration. All regimens will be given during patient hospitalization. A computer algorithm will be used in the randomization. The NPR was selected due to the expected significant anti-inflammatory activity and favorable cardiovascular safety profile.

All patients will be treated by the same surgical and anesthesiology team . Every effort will be made to follow the selection criteria recommended by the manufacturer of the stent graft, however, the surgeon' s decision as to which device to use will be based on the anatomical characteristics of the proximal neck, the iliac artery configuration, and the presence of thrombus or calcifications. Systemic heparinization will be achieved with 5,000 IU of heparin. Every effort will be made to deploy the endovascular device just below the level of the lowest renal artery. All the devices will be bifurcated systems. All patients will receive antibiotic prophylaxis (Daptomycin 500mg and Piperacillin/Tazobactam 2/0.25 gr) half an hour pre-operatively and for the day of operation, as well as 3500 IU of low molecular weight heparin (tinzaparin) from the first postoperative day until discharge.

In all patients, demographics, intra-operative and post-operative complications, the incidence of PIS, the diameter of the aneurysm, the type of the graft deployed, the operation time, the amount of contrast media administered and length of postoperative stay, will be recorded. Temperature will be recorded eight times daily for the duration of hospitalization. Blood tests including troponin levels will be measured on the first and second post-operative day and the day before discharge. Post-operative pain will be controlled with intravenous tramadol, while in cases of fever > 38.5oC lasting more than 2 hours intravenous paracetamol ( 1 g ) will be administered. All patients presenting with fever during the post-operative period, whether or not fulfilling the PIS criteria, will undergo a thorough work up for possible infection. If any of these tests reveal evidence of an early pulmonary, urinary tract or any other kind of infection, the patient will not be considered to suffer from PIS. Patients will be discharged in the absence of any complications, with a body temperature < 38oC for at least 24 hours and a WBC < 12.000/mL. Outpatient follow-up will be performed at 1, and 12 months after surgery.

Adverse events will include any major adverse cardiovascular events ( MACE ), acute renal failure, readmission, and death by any cause. MACE is defined as a composite of death from cardiac causes, non-fatal acute myocardial infarction ( ST and non-ST ), ischemic stroke, or transient ischemic attack. Death is considered due to cardiac causes if the patient died of MI, cardiac arrhythmia, or congestive heart failure caused primarily by a cardiac condition. The diagnosis of MI requires elevated troponin concentration with at least one of two 12-lead electrocardiogram changes, including development of new Q waves or new persistent ST-T segment or T wave changes.13 Unstable angina is defined as severe chest pain lasting for at least 30 minutes, unresponsive to standard therapeutic intervention, and associated with transient ST segment deviation of 0.05 mV, new or T wave inversion of 0.3 mV, without development of Q waves, or creatinine kinase-MB elevation. Stroke is defined according to the current World Health Organization definition as rapidly developing clinical signs of focal (or global) disturbance of cerebral function, lasting >24 hours or leading to death, with no apparent cause other than that of a vascular origin. Transient ischemic attack includes brief episodes of neurologic dysfunction resulting from focal cerebral ischemia, not associated with a permanent cerebral infarction, lasting < 24 hours. Acute kidney failure is defined as impaired renal function according to the Kidney Disease Improving Global Outcomes clinical practice guidelines.

All patients will be on antiplatelet therapy (aspirin 100 mg once daily) for at least 3 weeks prior to the procedure. Preoperative medications will be continued immediately after surgery. Patients who will become enrolled and will be already receiving a statin will continue their medication. For patients not already on statin, atorvastatin ( 20 mg once daily ) will be initiated at the screening visit.

Venous blood will be collected without a tourniquet preoperatively, at days 1 and 2 postoperatively. Besides the traditional inflammatory markers (WBC, hs-CRP, and fibrinogen ) interleukin 6 (IL-6) will be evaluated as it was the only marker significantly altered in PIS patients in a previous study.

STATISTICAL ANALYSIS Power analysis: Assuming the frequency of PIS after elective EVAR with a polyester endograft is 50%, the study will required 186 patients in both groups to have the 80 % power to detect a decrease in frequency to 30%.

Data will be expressed as mean ± standard deviation ( SD ) as appropriate, except for non-Gaussian parameters, which are presented as median (range). Comparisons of continuous variables will be performed by Student t test for normally distributed variables and Mann- Whitney U test for non-normally distributed variables, while the chi-square test was used for categorical variables. To assess the effect of the independent variables observed within the study context, each one will be initially examined separately and the significant predictors at level p1=.25 will be identified. These will be used in a binary logistic regression model. The formerly non-significant factors will then be considered again at level p2=.10. Interactions between the main effects of the final model will then be examined. The enter method with significance level p3=.05 will be used to obtain p values and odds ratios for the main effects and interactions. All analyses will be carried out with SPSS 20.0 statistical package for Windows (IBM Corporation, Armonk, New York).

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from infrarenal abdominal aortic aneurysm undergoing endovascular aneurysm repair

Exclusion Criteria:

* Leukocytosis (white blood cell count [WBC]> 10,000 / mL) and elevated body temperature

  * Signs of gangrene
  * Previous trauma or surgery two months before enrolling in the study
  * Previous implantation of endoprothesis
  * Any autoimmune disease or systemic inflammatory condition
  * Any malignancy
  * Use of anti-inflammatory drugs, chemotherapeutic agents, immunosuppressants or anticoagulants
  * Severe severe renal impairment (GFR < 30 ml / min) and
  * Absolute contraindications of NSAIDs such as: NSAID-allergic patients, patients who have experienced asthma attacks following the use of acetylsalicylic acid or other anti-inflammatory nonsteroidal drugs, patients with nasal polyps, patients with anaphylactic or other severe NSAID allergies, severe hepatic insufficiency, heart failure patients (moderate to severe), patients with ischemic heart disease or other vascular diseases, presence of old or active gastric or ulcer of duodenum, history of gastrointestinal haemorrhage in the past, proctitis or recent rectal bleeding, a history of inflammatory bowel disease (ulcerative colitis, Crohn's disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
major cardiovascular events after endovascular aneurysm repair | 2 years
  The occurrence of major cardiovascular event (myocardial infarction, stroke, transient ischemic attacks, cardiac arrythmia, congestive heart failure, angina unstable, cardiac death) after EVAR

SECONDARY OUTCOMES:
post implantation syndrome | 2 years
  the occurence of postimplantation syndrome after EVAR

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arnaoutoglou E, Papas N, Milionis H, Kouvelos G, Koulouras V, Matsagkas MI. Post-implantation syndrome after endovascular repair of aortic aneurysms: need for postdischarge surveillance. Interact Cardiovasc Thorac Surg. 2010 Oct;11(4):449-54. doi: 10.1510/icvts.2010.242628. Epub 2010 Jul 19. PMID 20643821
- [Result] Arnaoutoglou E, Kouvelos G, Milionis H, Mavridis A, Kolaitis N, Papa N, Papadopoulos G, Matsagkas M. Post-implantation syndrome following endovascular abdominal aortic aneurysm repair: preliminary data. Interact Cardiovasc Thorac Surg. 2011 Apr;12(4):609-14. doi: 10.1510/icvts.2010.256784. Epub 2011 Jan 19. PMID 21248083
- [Result] Arnaoutoglou E, Kouvelos G, Papa N, Kallinteri A, Milionis H, Koulouras V, Matsagkas M. Prospective evaluation of post-implantation inflammatory response after EVAR for AAA: influence on patients' 30 day outcome. Eur J Vasc Endovasc Surg. 2015 Feb;49(2):175-83. doi: 10.1016/j.ejvs.2014.12.006. Epub 2015 Jan 9. PMID 25579873
- [Result] Arnaoutoglou E, Kouvelos G, Papa N, Gartzonika K, Milionis H, Koulouras V, Matsagkas M. Prospective evaluation of postimplantation syndrome evolution on patient outcomes after endovascular aneurysm repair for abdominal aortic aneurysm. J Vasc Surg. 2016 May;63(5):1248-55. doi: 10.1016/j.jvs.2015.11.043. Epub 2016 Feb 28. PMID 26926930